CLINICAL TRIAL: NCT01836029
Title: A Randomized, Double-Blind, Placebo-Controlled Study of Chemotherapy Plus Cetuximab in Combination With VTX 2337 in Patients With Recurrent or Metastatic Squamous Cell Carcinoma of the Head and Neck
Brief Title: Chemotherapy Plus Cetuximab in Combination With VTX-2337 in Patients With Recurrent or Metastatic Squamous Cell Carcinoma of the Head and Neck
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VRXP-A202
Record Dates: First submitted 2013-04-12; First posted 2013-04-19 (Estimated); Results first posted 2019-10-29 (Actual); Last update posted 2019-10-29 (Actual); Status verified 2019-10

CONDITIONS: Carcinoma, Squamous Cell of Head and Neck
Keywords: SCCHN; HNSCC
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — VTX-2337; Carboplatin; Cisplatin; Fluorouracil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- chemotherapy and cetuximab plus VTX-2337 (Experimental): VTX-2337 (3.0 mg/m2) will be administered on Day 8 and Day 15 of a 21-day cycle for 6 cycles, followed by dosing on Days 8 and 22 of 28-day cycles until disease progression.
  Cisplatin (100 mg/m2) OR carboplatin (AUC 5 mg/mL/min) will be administered on Day 1 of a 21-day cycle for a maximum of 6 cycles.
  5-FU (1000 mg/m2) will be administered on Days 1-4 of a 21-day cycle for a maximum of 6 cycles.
  Cetuximab (initial dose: 400 mg/m2; remaining doses: 250 mg/m2) will be administered weekly until disease progression.
  Interventions: Drug: VTX-2337; Drug: Carboplatin; Drug: Cisplatin; Drug: 5-fluorouracil
- chemotherapy and cetuximab plus placebo (Active Comparator): Placebo (3.0 mg/m2) will be administered on Day 8 and Day 15 of a 21-day cycle for 6 cycles, followed by dosing on Days 8 and 22 of 28-day cycles until disease progression.
  Cisplatin (100 mg/m2) OR carboplatin (AUC 5 mg/mL/min) will be administered on Day 1 of a 21-day cycle for a maximum of 6 cycles.
  5-FU (1000 mg/m2) will be administered on Days 1-4 of a 21-day cycle for a maximum of 6 cycles.
  Cetuximab (initial dose: 400 mg/m2; remaining doses: 250 mg/m2) will be administered weekly until disease progression.
  Interventions: Drug: Carboplatin; Drug: Cisplatin; Drug: 5-fluorouracil; Drug: Placebo

INTERVENTIONS:
Drug: VTX-2337 — TLR8 Agonist
  Arms: chemotherapy and cetuximab plus VTX-2337
Drug: Carboplatin
  Other Names: paraplatin
Drug: Cisplatin
  Other Names: Platin
Drug: 5-fluorouracil
  Other Names: 5-FU; Efudex; Fluorouracil
Drug: Placebo
  Arms: chemotherapy and cetuximab plus placebo

SUMMARY:
The purpose of this study is to compare the progression-free survival of patients with recurrent or metastatic squamous cell carcinoma of the head and neck (SCCHN) treated with VTX-2337 + cisplatin or carboplatin + 5-FU + cetuximab versus patients treated with cisplatin or carboplatin + 5-FU + cetuximab alone (standard-of-care; SOC). Safety and overall survival will also be evaluated.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled, parallel group study to evaluate the safety and efficacy of VTX 2337 in combination with cisplatin or carboplatin, 5-FU and cetuximab in prolonging the progression-free survival in subjects with recurrent or metastatic squamous cell carcinoma of the head and neck.

OBJECTIVES:

Primary Objective:

To compare the efficacy of VTX 2337 plus SOC to SOC alone in prolonging the PFS of patients with recurrent or metastatic SCCHN using irRECIST evaluated by independent radiology review.

Secondary Objectives:

To compare the following between the two treatment groups:

* Safety of VTX 2337 by adverse events, including clinically significant changes in physical examination, peripheral blood hematology, serum chemistry, urinalysis, and ECG.
* Efficacy of VTX 2337 plus SOC in prolonging the OS of patients with recurrent or metastatic SCCHN.
* Efficacy of VTX-2337 plus SOC on ORR, DOBR, DCR, and DDC by irRECIST and evaluation by independent radiology review.
* Efficacy of VTX-2337 plus SOC on ORR, DOBR, DCR, and DDC by RECIST v1.1 and evaluation by independent radiology review.
* Efficacy of VTX 2337 plus SOC to SOC alone in prolonging the PFS by RECIST v1.1 and evaluation by independent radiology review.
* Efficacy of VTX 2337 plus SOC to SOC alone in prolonging the PFS by irRECIST and evaluation by investigators.

Exploratory Objectives:

* To compare genetic polymorphisms that may impact the response of patients to a TLR8 agonist or to cetuximab between the two treatment groups.
* To compare immune biomarker response to VTX 2337 plus SOC as measured by a multiplexed panel of cytokines, chemokines, and inflammatory markers between the two treatment groups.
* To compare the effect of immune cell subsets within the tumor on response to VTX-2337 and/or clinical outcome, as measured by immunohistochemistry in primary tumor tissue between the two treatment groups.
* To assess the PK of VTX-2337.

OUTLINE:

Subjects will be screened for eligibility (within 14 days) and qualified subjects will be randomized 1:1 to 1 of 2 treatment groups: SOC + VTX 2337 or SOC + placebo.

Tumor assessments will be by CT or MRI starting at Week 12 (± 3 days), then at Week 18 (± 3 days) and every 8 weeks (± 7 days) thereafter. Response will be evaluated by immune-related RECIST criteria (irRECIST) and confirmed by an independent radiologist.

Upon independent confirmation of disease progression, active participation in the study is complete and subjects will undergo the End of Treatment evaluations.

Subjects will be followed for survival until ~12 months after the last subject is randomized.

ELIGIBILITY:
Inclusion Criteria:

* Ability and willingness to provide written informed consent
* Histologically or cytologically confirmed squamous cell carcinoma of the head and neck
* Locoregionally recurrent or metastatic disease that has not previously been treated with systemic therapy of recurrent or metastatic disease
* At least one measurable lesion on screening CT or MRI
* 18 years of age or older
* ECOG performance status of 0 or 1
* Acceptable bone marrow, renal, and hepatic function based upon screening lab tests
* Willingness to use medically acceptable contraception
* For females with reproductive potential: a negative serum pregnancy test

Exclusion Criteria:

* Disease which is amenable to curative local therapy
* Nasopharyngeal, salivary gland, lip or sinonasal carcinoma
* Surgery or irradiation ≤ 4 weeks prior to randomization
* Prior systemic anti-cancer therapy, unless administered for localized SCCHN and completed at least 6 months prior to disease recurrence
* Treatment with an investigational agent ≤ 30 days prior to randomization
* Treatment with corticosteroids within 2 weeks
* A requirement for chronic systemic immunosuppressive therapy for any reason
* Prior serious infusion reaction to cetuximab
* Treatment with an immunotherapy within 30 days
* Known brain metastases, unless stable for at least 28 days
* Active autoimmune disease currently requiring therapy
* Known infection with HIV
* Significant cardiac disease within 6 months
* Pregnant or breast-feeding females
* History of another primary malignancy, with the exception of (i) curatively resected non-melanoma skin cancer, (ii) curatively treated in situ cervical cancer, or (iii) other malignancy curatively treated with no evidence of disease and no anticancer therapy administered for 3 years prior to randomization, with the exception of adjuvant hormonal therapy for breast cancer
* Other conditions or circumstances that could interfere with the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 195 (Actual)
Dates: Start 2013-10-14 (Actual); Primary Completion 2016-04-13 (Actual); Study Completion 2016-09-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ezra Cohen, MD, Study Chair — University of Chicago; Robert Ferris, MD, PhD, Study Chair — University of Pittsburgh; Amar Patel, MD, Study Director — Celgene
Locations (53):
- United States (53):
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Tower Hematology Oncology Medical Group, Beverly Hills, California
  - California Cancer Associates for Research and Excellence (CCARE), Escondido, California
  - University of California San Diego Moores Cancer Center, La Jolla, California
  - University of California Norris Comprehensive Cancer Center, Los Angeles, California
  - University of Colorado Cancer Center, Aurora, Colorado
  - VA Eastern Colorado Healthcare System, Denver, Colorado
  - Helen F. Graham Cancer Center, Newark, Delaware
  - MD Anderson Cancer Center, Orlando, Florida
  - Northeast Georgia Cancer Care, LLC, Athens, Georgia
  - Winship Cancer Institute, Atlanta, Georgia
  - Tripler Army Medical Center, Honolulu, Hawaii
  - Northwestern University Feinberg School of Medicine, Chicago, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - University of Kansas Cancer Center, Westwood, Kansas
  - Crescent City Research Consortium, LLC, Marrero, Louisiana
  - Robert W. Veith, MD, LLC, Metairie, Louisiana
  - Maine Center for Cancer Medicine, Scarborough, Maine
  - The Sidney Kimmel Comprehensive Cancer Center at John Hopkins, Baltimore, Maryland
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Health System, Detroit, Michigan
  - Providence Cancer Institute, Southfield, Michigan
  - Saint Louis Cancer Care, LLP, Bridgeton, Missouri
  - Barnes Jewish Hospital, St Louis, Missouri
  - Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Oncology and Hematology Specialists, P.A., Denville, New Jersey
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Monter Cancer Center, Lake Success, New York
  - The Bellevue Hospital, New York, New York
  - Mount Sinai Medical Center, New York, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Wake Forest University Baptist Medical Center, Winston-Salem, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - University Hospitals of Cleveland, Cleveland, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Saint Charles Medical Center, Bend, Oregon
  - Providence Cancer Center, Portland, Oregon
  - Saint Lukes Cancer Centre, Easton, Pennsylvania
  - Pennsylvania State Hershey Cancer Institute, Hershey, Pennsylvania
  - University of Pittsburgh Cancer Institute, Pittsburgh, Pennsylvania
  - Hollings Cancer Center, Charleston, South Carolina
  - The West Clinic, Memphis, Tennessee
  - University of Texas Southwestern Medical Center at Dallas, Dallas, Texas
  - San Antonio Military Medical Center, Fort Sam Houston, Texas
  - Virginia Cancer Specialists, PD, Fairfax, Virginia
  - Medical Oncology Associates, PS, Spokane, Washington
  - Madigan Army Medical Center, Tacoma, Washington
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Aurora Advanced Healthcare, Inc., Wauwatosa, Wisconsin

REFERENCES:
- [Derived] Ferris RL, Saba NF, Gitlitz BJ, Haddad R, Sukari A, Neupane P, Morris JC, Misiukiewicz K, Bauman JE, Fenton M, Jimeno A, Adkins DR, Schneider CJ, Sacco AG, Shirai K, Bowles DW, Gibson M, Nwizu T, Gottardo R, Manjarrez KL, Dietsch GN, Bryan JK, Hershberg RM, Cohen EEW. Effect of Adding Motolimod to Standard Combination Chemotherapy and Cetuximab Treatment of Patients With Squamous Cell Carcinoma of the Head and Neck: The Active8 Randomized Clinical Trial. JAMA Oncol. 2018 Nov 1;4(11):1583-1588. doi: 10.1001/jamaoncol.2018.1888. PMID 29931076
- [Derived] Chow LQM, Morishima C, Eaton KD, Baik CS, Goulart BH, Anderson LN, Manjarrez KL, Dietsch GN, Bryan JK, Hershberg RM, Disis ML, Martins RG. Phase Ib Trial of the Toll-like Receptor 8 Agonist, Motolimod (VTX-2337), Combined with Cetuximab in Patients with Recurrent or Metastatic SCCHN. Clin Cancer Res. 2017 May 15;23(10):2442-2450. doi: 10.1158/1078-0432.CCR-16-1934. Epub 2016 Nov 3. PMID 27810904
- [Derived] Northfelt DW, Ramanathan RK, Cohen PA, Von Hoff DD, Weiss GJ, Dietsch GN, Manjarrez KL, Randall TD, Hershberg RM. A phase I dose-finding study of the novel Toll-like receptor 8 agonist VTX-2337 in adult subjects with advanced solid tumors or lymphoma. Clin Cancer Res. 2014 Jul 15;20(14):3683-91. doi: 10.1158/1078-0432.CCR-14-0392. Epub 2014 May 7. PMID 24807889

RESULTS

PARTICIPANT FLOW:
Groups:
- Chemotherapy and Cetuximab Plus VTX-2337: VTX-2337 (3.0 mg/m2) will be administered on Day 8 and Day 15 of a 21-day cycle for 6 cycles, followed by dosing on Days 8 and 22 of 28-day cycles until disease progression. Cisplatin (100 mg/m2) OR carboplatin (AUC 5 mg/mL/min) will be administered on Day 1 of a 21-day cycle for a maximum of 6 cycles. 5-FU (1000 mg/m2) will be administered on Days 1-4 of a 21-day cycle for a maximum of 6 cycles. Cetuximab (initial dose: 400 mg/m2; remaining doses: 250 mg/m2) will be administered weekly until disease progression. VTX-2337: TLR8 Agonist Carboplatin Cisplatin 5-fluorouracil
- Chemotherapy and Cetuximab Plus Placebo: Placebo (3.0 mg/m2) will be administered on Day 8 and Day 15 of a 21-day cycle for 6 cycles, followed by dosing on Days 8 and 22 of 28-day cycles until disease progression. Cisplatin (100 mg/m2) OR carboplatin (AUC 5 mg/mL/min) will be administered on Day 1 of a 21-day cycle for a maximum of 6 cycles. 5-FU (1000 mg/m2) will be administered on Days 1-4 of a 21-day cycle for a maximum of 6 cycles. Cetuximab (initial dose: 400 mg/m2; remaining doses: 250 mg/m2) will be administered weekly until disease progression. Carboplatin Cisplatin 5-fluorouracil Placebo
Period: Overall Study
Arm/Group | Chemotherapy and Cetuximab Plus VTX-2337 | Chemotherapy and Cetuximab Plus Placebo
Started | 100 | 95
Completed | 100 | 95
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Chemotherapy and Cetuximab Plus VTX-2337 | Chemotherapy and Cetuximab Plus Placebo | Total
Number analyzed (Participants) | 100 | 95 | 195
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.1 (10.07) | 59.9 (9.08) | 58.5 (9.68)
Age, Customized [Count of Participants; unit: Participants]
  <40 years | 6 | 1 | 7
  40-49 years | 9 | 9 | 18
  50-59 years | 47 | 35 | 82
  60-69 years | 29 | 37 | 66
  70-79 years | 8 | 13 | 21
  >=80 years | 1 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 14 | 29
  Male | 85 | 81 | 166
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 15 | 12 | 27
  White | 81 | 78 | 159
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 3 | 6
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 100 | 95 | 195

OUTCOME MEASURES:

1. Primary Outcome: Comparison of Progression Free Survival (PFS) Between Treatment Groups Using irRECIST and Evaluated by Independent Radiology.
Description: PFS was based on central assessment by a blinded independent radiologist per immune related response evaluation criteria for solid tumors (irRECIST) and was summarized and displayed by treatment arm using Kaplan-Meier methods. Treatments were compared using a stratified log-rank test controlling for randomization stratification factors. The hazard ratio between the 2 treatment arms, as well as the associated one-sided 90% CI and p-value, were presented using a Cox proportional hazards regression model.
Time Frame: PFS is the time from randomization until disease progression or death, whichever comes first.
Population: ITT population
Measure: Median (90% Confidence Interval); unit: days
Arm/Group | Chemotherapy and Cetuximab Plus VTX-2337 | Chemotherapy and Cetuximab Plus Placebo
Number analyzed (Participants) | 100 | 95
days | 185 [182 to NA] — The upper bound of the confidence interval could not be calculated. | 181 [180 to NA] — The upper bound of the confidence interval could not be calculated.
Statistical Analysis 1: Comparison: Chemotherapy and Cetuximab Plus VTX-2337 vs Chemotherapy and Cetuximab Plus Placebo; Test type: Superiority or Other; p = 0.266, Log Rank — The 1-sided p-value based on a log-rank test stratified by randomization stratification factors; Hazard Ratio (HR) = 0.99, 90% CI 1-sided [upper limit 1.22]

2. Secondary Outcome: Comparison of Adverse Events (AEs) Between the Two Treatment Groups.
Description: The frequency and severity of adverse events, including any clinically significant changes in physical exam, laboratory values, or other clinical assessment.
Time Frame: AEs were collected from the first dose of study drug given on Cycle 1 Day 1 until 7 days after the dose of study drug or End of Treatment visit, whichever occurred first. Overall mean duration of exposure was 25.3 weeks.
Population: Safety population: subjects who received at least 1 dose of VTX-2337 or placebo.
Measure: Number; unit: percentage of participants
Arm/Group | Chemotherapy and Cetuximab Plus VTX-2337 | Chemotherapy and Cetuximab Plus Placebo
Number analyzed (Participants) | 89 | 86
percentage of participants
  Subjects with TEAE | 100 | 100
  Subjects with Grade 3 and above TEAE | 84.3 | 83.7
  Subjects with serious TEAE | 39.3 | 39.5
  Subjects with TEAE with outcome of death | 4.5 | 8.1
  Subjects discontinued treatment due to TEAE | 19.1 | 18.6

3. Secondary Outcome: Comparison of Overall Survival (OS) Between the 2 Treatment Groups.
Description: Estimated using Kaplan-Meier product limit estimates, 1-sided stratified log-rank test, and Cox proportional hazard model; all with 90% 1-sided confidence intervals.
Time Frame: OS is the time from randomization until death due to any cause or the date last confirmed to be alive.
Population: ITT population
Measure: Median (90% Confidence Interval); unit: days
Arm/Group | Chemotherapy and Cetuximab Plus VTX-2337 | Chemotherapy and Cetuximab Plus Placebo
Number analyzed (Participants) | 100 | 95
days | 412 [359 to NA] — The upper bound of the confidence interval could not be calculated. | 343 [319 to NA] — The upper bound of the confidence interval could not be calculated.
Statistical Analysis 1: Comparison: Chemotherapy and Cetuximab Plus VTX-2337 vs Chemotherapy and Cetuximab Plus Placebo; Test type: Superiority or Other; p = 0.399, Log Rank — The 1-sided p-value based on a log-rank test stratified by randomization stratification factors; Hazard Ratio (HR) = 0.95, 90% CI 1-sided [upper limit 1.22]

4. Secondary Outcome: Comparison of the Objective Response Rate Between the Two Treatment Groups p
Description: Objective response rate is defined as the percentage of subjects who achieve best overall response of irCR or irPR pr irRECIST and evaluated by independent radiology..
Time Frame: From the time of randomization until the best response on treatment is documented.
Population: ITT population
Measure: Number; unit: percentage of participants
Arm/Group | Chemotherapy and Cetuximab Plus VTX-2337 | Chemotherapy and Cetuximab Plus Placebo
Number analyzed (Participants) | 100 | 95
percentage of participants | 38.0 | 33.7
Statistical Analysis 1: Comparison: Chemotherapy and Cetuximab Plus VTX-2337 vs Chemotherapy and Cetuximab Plus Placebo; Test type: Superiority or Other; p = 0.536, Cochran-Mantel-Haenszel — p-values are from Cochran-Mantel-Haenszel tests controlling for randomization stratification factors and comparing tumor response rates between the treatment groups

ADVERSE EVENTS:
Time Frame: AE data was collected from the first patient's Cycle 1 Day 1, 14 Oct 2013, through primary analysis data cut date, 13 Apr 2016. AEs were collected from the first dose of study drug given on Cycle 1 Day 1 until 7 days after the dose of study drug or End of Treatment visit, whichever occurred first. The whole period equals to 2.5 years.
Description: AEs were collected through reporting voluntarily by the subject, discovery via questioning by the investigator or clinical personnel, or identification through physical examination, laboratory test or other means. Overall mean duration of exposure was 25.3 weeks for study drug.
Arm/Group | Chemotherapy and Cetuximab Plus VTX-2337 | Chemotherapy and Cetuximab Plus Placebo
Serious Adverse Events (participants affected / at risk) | 35/89 | 34/86
Other Adverse Events (participants affected / at risk) | 89/89 | 86/86
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Chemotherapy and Cetuximab Plus VTX-2337 (N=89) | Chemotherapy and Cetuximab Plus Placebo (N=86)
Pneumonia (Infections and infestations) | 5 | 5
Neutropenia (Blood and lymphatic system disorders) | 7 | 2
Dehydration (Metabolism and nutrition disorders) | 5 | 4
vomitting (Gastrointestinal disorders) | 5 | 3
Nausea (Gastrointestinal disorders) | 4 | 2
Sepsis (Infections and infestations) | 2 | 4
Lung infection (Infections and infestations) | 3 | 1
Pulmonary emolism (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Hypotension (Vascular disorders) | 1 | 4
Fatigue (General disorders) | 2 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Anaemia (Blood and lymphatic system disorders) | 3 | 0
Pancytopenia (Blood and lymphatic system disorders) | 1 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 1
Cardiac arrest (Cardiac disorders) | 0 | 2
Leukopenia (Blood and lymphatic system disorders) | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 3 | 4
Acute coronary syndrome (Cardiac disorders) | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 0
Atrioventricular block second degree (Cardiac disorders) | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 1 | 0
Palpitations (Cardiac disorders) | 1 | 0
Pericarditis (Cardiac disorders) | 0 | 1
Sinus tachycardia (Cardiac disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 1
Dysphagia (Gastrointestinal disorders) | 1 | 1
Enterocolitis (Gastrointestinal disorders) | 0 | 1
Haematemesis (Gastrointestinal disorders) | 1 | 0
Ileus (Gastrointestinal disorders) | 0 | 1
Melaena (Gastrointestinal disorders) | 1 | 0
Mouth haemorrhage (Gastrointestinal disorders) | 1 | 0
Oesophageal perforation (Gastrointestinal disorders) | 0 | 1
Pneumatosis intestinalis (Gastrointestinal disorders) | 0 | 1
Pneumoperitoneum (Gastrointestinal disorders) | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 2
Asthenia (General disorders) | 0 | 1
Death (General disorders) | 0 | 2
Medical device complication (General disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 0 | 1
Pain (General disorders) | 1 | 2
Pyrexia (General disorders) | 3 | 0
Anaphylactic reaction (Immune system disorders) | 1 | 1
Cytokine release syndrome (Immune system disorders) | 1 | 0
Hypersensitivity (Immune system disorders) | 0 | 1
Acinetobacter bacteraemia (Infections and infestations) | 0 | 1
Bacteraemia (Infections and infestations) | 1 | 1
Clostridium difficile infection (Infections and infestations) | 0 | 1
Device related infection (Infections and infestations) | 0 | 1
Infection (Infections and infestations) | 1 | 0
Neutropenic sepsis (Infections and infestations) | 0 | 2
Pneumonia bacterial (Infections and infestations) | 0 | 1
Soft tissue infection (Infections and infestations) | 1 | 0
Staphylococcal infection (Infections and infestations) | 1 | 0
Staphylococcal sepsis (Infections and infestations) | 1 | 0
Tracheitis (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1
Feeding tube complication (Injury, poisoning and procedural complications) | 0 | 1
Forearm fracture (Injury, poisoning and procedural complications) | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 1 | 1
Radiation mucositis (Injury, poisoning and procedural complications) | 0 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 1
Occult blood positive (Investigations) | 1 | 0
Acidosis (Metabolism and nutrition disorders) | 0 | 1
Failure to thrive (Metabolism and nutrition disorders) | 0 | 2
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 0
Metabolic syndrome (Metabolism and nutrition disorders) | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 2
Convulsion (Nervous system disorders) | 0 | 1
Haemorrhage intracranial (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 1
Ischaemic stroke (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 0 | 2
Mental status changes (Psychiatric disorders) | 1 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 2
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Upper airway obstruction (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Swelling face (Skin and subcutaneous tissue disorders) | 1 | 0
Wound treatment (Surgical and medical procedures) | 0 | 1
Embolism (Vascular disorders) | 1 | 1
Shock haemorrhagic (Vascular disorders) | 0 | 1
Vena cava thrombosis (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Chemotherapy and Cetuximab Plus VTX-2337 (N=89) | Chemotherapy and Cetuximab Plus Placebo (N=86)
Anaemia (Blood and lymphatic system disorders) | 53 | 39
Leukopenia (Blood and lymphatic system disorders) | 38 | 29
Lymphopenia (Blood and lymphatic system disorders) | 10 | 9
Neutropenia (Blood and lymphatic system disorders) | 50 | 45
Thrombocytopenia (Blood and lymphatic system disorders) | 50 | 43
Tachycardia (Cardiac disorders) | 8 | 4
Constipation (Gastrointestinal disorders) | 30 | 23
Diarrhoea (Gastrointestinal disorders) | 28 | 26
Dry mouth (Gastrointestinal disorders) | 2 | 9
Dyspepsia (Gastrointestinal disorders) | 7 | 5
Dysphagia (Gastrointestinal disorders) | 11 | 15
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 | 7
Nausea (Gastrointestinal disorders) | 36 | 29
Oral pain (Gastrointestinal disorders) | 5 | 5
Stomatitis (Gastrointestinal disorders) | 34 | 42
Vomiting (Gastrointestinal disorders) | 32 | 24
Asthenia (General disorders) | 4 | 6
Chills (General disorders) | 33 | 5
Fatigue (General disorders) | 38 | 39
Influenza like illness (General disorders) | 13 | 3
Injection site reactions (General disorders) | 35 | 0
Pain (General disorders) | 4 | 6
Pyrexia (General disorders) | 38 | 10
Cytokine release syndrome (Immune system disorders) | 7 | 3
Paronychia (Infections and infestations) | 8 | 10
Pneumonia (Infections and infestations) | 8 | 7
Alanine aminotransferase increased (Investigations) | 3 | 8
Blood alkaline phosphatase increased (Investigations) | 8 | 9
Weight decreased (Investigations) | 24 | 26
Decreased appetite (Metabolism and nutrition disorders) | 22 | 15
Dehydration (Metabolism and nutrition disorders) | 15 | 19
Hyperglycaemia (Metabolism and nutrition disorders) | 11 | 8
Hypoalbuminaemia (Metabolism and nutrition disorders) | 14 | 9
Hypocalcaemia (Metabolism and nutrition disorders) | 9 | 10
Hypokalaemia (Metabolism and nutrition disorders) | 29 | 24
Hypomagnesaemia (Metabolism and nutrition disorders) | 26 | 31
Hyponatraemia (Metabolism and nutrition disorders) | 14 | 13
Arthralgia (Musculoskeletal and connective tissue disorders) | 12 | 6
Back pain (Musculoskeletal and connective tissue disorders) | 10 | 6
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 4 | 5
Neck pain (Musculoskeletal and connective tissue disorders) | 7 | 6
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 8
Dizziness (Nervous system disorders) | 13 | 20
Dysgeusia (Nervous system disorders) | 11 | 8
Headache (Nervous system disorders) | 10 | 13
Neuropathy peripheral (Nervous system disorders) | 9 | 10
Anxiety (Psychiatric disorders) | 6 | 7
Depression (Psychiatric disorders) | 8 | 6
Insomnia (Psychiatric disorders) | 5 | 8
Cough (Respiratory, thoracic and mediastinal disorders) | 15 | 16
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 3 | 7
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 8 | 14
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 8 | 4
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 5 | 5
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 7 | 8
Alopecia (Skin and subcutaneous tissue disorders) | 4 | 6
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 43 | 31
Dry skin (Skin and subcutaneous tissue disorders) | 10 | 20
Pruritus (Skin and subcutaneous tissue disorders) | 5 | 9
Rash (Skin and subcutaneous tissue disorders) | 17 | 23
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 9 | 5
Skin fissures (Skin and subcutaneous tissue disorders) | 12 | 20
Hypertension (Vascular disorders) | 4 | 5
Hypotension (Vascular disorders) | 4 | 15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI should not publish the site's results prior to the sponsor's 1st multi-site publication. PI can publish if no multi-site publication within 18 months after the study has been completed or terminated, provided that the site's results are statistically significant and consistent with the multi-site publication. Prior to submitting or presenting, PI should provide sponsor to review and comment. If requested by sponsor, PI should delay publication/presentation for up to 120 days.